CLINICAL TRIAL: NCT06197373
Title: Outcomes of Early and Late Laparoscopic Cholecystectomy (LC) After Endoscopic Retrograde CholangioPancreatography (ERCP), Prospective Study .
Brief Title: Laparoscopic Cholecystectomy After ERCP
Status: Not yet recruiting | Type: Observational
Sponsor: Mohamed Bakr Mohamed Ahmed (Other)
Responsible Party: Sponsor-Investigator, Mohamed Bakr Mohamed Ahmed, Head of general surgery at assuit university, Assiut University
Organization: Assiut University (Other)
Other Study IDs: cholecystectomy after ERCP
Record Dates: First submitted 2023-12-09; First posted 2024-01-09 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Laparoscopic Cholecystectomy
MeSH Terms: interventions — Cholecystectomy, Laparoscopic; Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 21 Days

GROUPS / COHORTS (2):
- Early laparoscopic cholecystectomy after ERCP: Evaluation of outcomes of early ( within 72 hours) laparoscopic cholecystectomy after ERCP
  Interventions: Procedure: Laparoscopic cholecystectomy
- Late laparoscopic cholecystectomy after ERCP: Evaluation of outcomes of late ( form third day up to 2months ) laparoscopic cholecystectomy after ERCP
  Interventions: Procedure: Laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy — Doing laparoscopic cholecystectomy after ERCP at different intervals
  Other Names: ERCP

SUMMARY:
Evaluation of outcomes of early and late laparoscopic cholecystectomy after ERCP

DETAILED DESCRIPTION:
Evaluation of both benefits and harms of doing laparoscopic cholecystectomy early within first 72 hours and late from the third day up to 2 months after ERCP

ELIGIBILITY:
Inclusion Criteria:

* female patient
* 18-60 years old

Exclusion Criteria:

* male patient
* extremes of age less than 18 and more than 60

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Female patient present with CBD obstruction and GB stones So Undergoing ERCP then Laparoscopic cholecystectomy
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Duration of the operation | 5 hours
  Measuring the time of the operation
Bleeding during operation | 5 hours
  Measuring amount of blood loss during operation
Hospital stay duration | 7 days
  Measuring time of hospital stay
Rate of Conversion to open cholecystectomy | 5 hours
  Documenting number of cases undergoing conversion from laparoscopic to open cholecystectomy

SECONDARY OUTCOMES:
Total cost of the medical service in both categories | 2 months
  Measuring the cost of the medical service in both categories for economic preference

CONTACTS AND LOCATIONS:
Overall Officials: Thabet, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided